CLINICAL TRIAL: NCT06420765
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Parallel Study Evaluating the Effects of Single Doses of NaV1.8 Inhibitors on C-Nociceptor Action Potentials in Healthy Adults
Brief Title: A Microneurography Study of NaV1.8 Inhibition in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VX23-PMI-001
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VX-150 (Experimental): Participants will be randomized to receive a single dose of VX-150.
  Interventions: Drug: VX-150
- VX-548 (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-548
  Interventions: Drug: VX-548
- VX-993 (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-993.
  Interventions: Drug: VX-993
- Placebo (Placebo Comparator): Participants will receive single dose of non-matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-150 — Suspension for oral administration.
  Arms: VX-150
Drug: VX-548 — Solution or suspension for oral administration.
  Arms: VX-548
Drug: VX-993 — Suspension for oral administration.
  Arms: VX-993
Drug: Placebo — Suspension for oral administration.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of Nav1.8 inhibition on activity-dependent slowing (ADS) of C-nociceptor nerve fibers, evoked action potential (AP) conduction velocity of C-nociceptor nerve fibers using VX-150, VX-993 and VX-548.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before study drug dosing
* Any condition possibly affecting drug absorption
* Any dermatological (generalized) or autoimmune disease that may affect C-nociceptor excitability
* Participants with Type 1 or Type 2 diabetes mellitus
* Participants who have any 1 of the following criteria in the foot in which microneurography (MNG) will be performed:

  * Injection of local anesthetics or steroids within 35 days prior to randomization.
  * Unsuitable anatomy of the superficial peroneal nerve (i.e., nerve cannot be seen or palpated at the dorsum of the foot)
  * Infection, disease (dermatologic or vascular), ongoing pain, or recent trauma or surgery that may affect study assessments Note: Participants must have 1 foot that does not meet any of the above criteria to be eligible.

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Activity Dependent Slowing (ADS) Over Time | From Pre-dose up to 2-hours Post Dose

SECONDARY OUTCOMES:
Change From Baseline in Conduction Velocity at 0.25 Hz Over Time | From Pre-dose up to 2-hours Post Dose
Change From Baseline in Action Potential (AP) Latency at 0.25 Hz Over Time | From Pre-dose up to 2-hours Post Dose
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAE) | From Day 1 up to Day 16

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing